CLINICAL TRIAL: NCT00036855
Title: A Phase I Study Of Yttrium-Ibritumomab Tiuxetan (90Y Zevalin, Yttrium (90)-Anti-CD20, NSC # 710085) Preceded By Rituximab In Children With Recurrent/Refractory CD20 Positive Lymphoma
Brief Title: Radiolabeled Monoclonal Antibody With or Without Peripheral Stem Cell Transplantation in Treating Children With Recurrent or Refractory Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01871; ADVL0013; U01CA097452 (NIH); CDR0000069331 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-05-13; First posted 2003-01-27 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: AIDS-related Peripheral/Systemic Lymphoma; AIDS-related Primary CNS Lymphoma; Post-transplant Lymphoproliferative Disorder; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent/Refractory Childhood Hodgkin Lymphoma
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating; Burkitt Lymphoma; Recurrence | interventions — Rituximab; Indium; ibritumomab tiuxetan; Peripheral Blood Stem Cell Transplantation; Filgrastim; Granulocyte Colony-Stimulating Factor

ARMS (2):
- Group A (no planned PBSC support) (Experimental): Patients receive rituximab IV over 4-6 hours followed by IDEC-In2B8 IV over 10 minutes on day 0 and undergo whole body imaging. Patients may then receive rituximab IV over 4-6 hours followed by IDEC-Y2B8 IV over 10 minutes on day 7.
  Some patients receive autologous PBSC IV over 30-60 minutes on day 35.
  Interventions: Biological: rituximab; Radiation: indium In 111 ibritumomab tiuxetan; Radiation: yttrium Y 90 ibritumomab tiuxetan; Procedure: peripheral blood stem cell transplantation; Other: laboratory biomarker analysis
- Group B (planned PBSC support) (Experimental): Patients receive rituximab, IDEC-In2B8, and IDEC-Y2B8 as in group A. Patients also receive autologous PBSC IV over 30-60 minutes on day 21 and G-CSF subcutaneously beginning on day 22 and continuing until blood counts recover or day 35.
  Interventions: Biological: rituximab; Radiation: indium In 111 ibritumomab tiuxetan; Radiation: yttrium Y 90 ibritumomab tiuxetan; Procedure: peripheral blood stem cell transplantation; Biological: filgrastim; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Radiation: indium In 111 ibritumomab tiuxetan — Given IV
  Other Names: IDEC-In2B8
Radiation: yttrium Y 90 ibritumomab tiuxetan — Given IV
  Other Names: 90Y ibritumomab tiuxetan; IDEC Y2B8; Y90 Zevalin; Y90-labeled ibritumomab tiuxetan
Procedure: peripheral blood stem cell transplantation — Undergo PBSC transplantation
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Biological: filgrastim — Given subcutaneously
  Other Names: G-CSF; Neupogen
  Arms: Group B (planned PBSC support)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase I trial to study the effectiveness of radiolabeled monoclonal antibody therapy with or without peripheral stem cell transplantation in treating patients who have recurrent or refractory lymphoma. Radiolabeled monoclonal antibodies can locate cancer cells and deliver radioactive tumor-killing substances to them without harming normal cells. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by anticancer therapy

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of yttrium Y 90 ibritumomab tiuxetan (IDEC-Y2B8) when preceded by rituximab in children with recurrent or refractory CD20-positive lymphoma for which no autologous peripheral blood stem cell transplantation (AuPBSCT) is planned. (Group A) If the dose-limiting toxicity (DLT) in group A is purely hematological, determine the MTD of IDEC-Y2B8 when combined with rituximab, AuPBSCT, and filgrastim (G-CSF) in a second group of children with recurrent or refractory CD20-positive lymphoma. (Group B) II. Determine the DLT of rituximab and IDEC-Y2B8 in these patients. III. Determine the dosimetry of indium In 111 ibritumomab tiuxetan preceded by rituximab in these patients.

IV. Determine, preliminarily, the antitumor activity of rituximab and IDEC-Y2B8 in these patients.

V. Assess the immune cell depletion (B-cell and T-cell) and recovery in patients treated with this regimen.

VI. Determine the human anti-mouse antibody response in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of yttrium Y 90 ibritumomab tiuxetan (IDEC-Y2B8). Patients are assigned to 1 of 2 groups.

GROUP A (no planned peripheral blood stem cell [PBSC] support): Patients receive rituximab IV over 4-6 hours followed by indium In 111 ibritumomab tiuxetan (IDEC-In2B8) IV over 10 minutes on day 0 and undergo whole body imaging. Patients may then receive rituximab IV over 4-6 hours followed by IDEC-Y2B8 IV over 10 minutes on day 7.

Cohorts of 3-6 patients in each subgroup (A1, A2, and A3) receive escalating doses of IDEC-Y2B8 until the maximum tolerated dose (MTD) is determined (subgroup A1 closed as of 10/8/04). The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity (DLT).

Some patients receive autologous PBSC IV over 30-60 minutes on day 35.

GROUP B (planned PBSC support): Patients receive rituximab, IDEC-In2B8, and IDEC-Y2B8 as in group A. Patients also receive autologous PBSC IV over 30-60 minutes on day 21 and filgrastim (G-CSF) subcutaneously beginning on day 22 and continuing until blood counts recover or day 35.

If the DLT in group A is purely hematological, cohorts of 3-6 patients in group B receive escalating doses of IDEC-Y2B8 until the MTD is determined. The MTD is defined as in group A.

Patients in both groups are followed at days 63, 90, 180, 365, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed and immunophenotypically (CD20)-positive lymphoma at original diagnosis, progression, or relapse
* Refractory to conventional therapy

  * First recurrent/refractory CD20-positive non-Hodgkin's lymphoma (NHL) allowed if ineligible for or refused regimens with known curative potential (high-dose chemotherapy plus bone marrow transplantation) (if available)
  * Second or third progression and/or recurrence of NHL
  * Second or third relapse/refractory CD20-positive Hodgkin's lymphoma
  * CD20-positive, post-transplantation lymphoproliferative lymphoma that is medically refractory (decreased immunosuppression) to rituximab and/or chemotherapy
  * Medically refractory, HIV-associated, CD20-positive NHL
  * Recurrent/refractory CD20-positive lymphoblastic lymphoma
* Autologous peripheral blood stem cells (PBSC) collected, selected for a minimum of 2 x 10^6 CD34-positive cells per kg, and cryopreserved before study entry
* Meets one of the following criteria for bone marrow reserve:

  * Good marrow reserve, defined by both of the following:

    * No prior myeloablative stem cell transplantation (SCT)
    * No prior extensive radiotherapy, defined by any of the following:

      * Prior total body irradiation
      * Prior radiotherapy dose of 3,600 cGy or more to cranio-spinal axis
      * Prior radiotherapy to 50% or more of bone marrow
  * Poor marrow reserve, defined by either or both of the following:

    * Prior myeloablative SCT
    * Prior extensive radiotherapy
* Performance status - Lansky 50-100% (age 10 and under)
* Performance status - Karnofsky 50-100% (age 11 to 21)
* At least 2 months
* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3 for patients with poor marrow reserve (transfusion independent)
* Platelet count ≥ 150,000 for patients with good marrow reserve (transfusion independent)
* Hemoglobin ≥ 8.0 g/dL (transfusion allowed)
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT ≤ 5 times ULN
* Albumin ≥ 2 g/dL
* Creatinine normal
* Creatinine clearance or glomerular filtration rate ≥ 70 mL/min
* Shortening fraction ≥ 27% by echocardiogram
* Ejection fraction ≥ 50% by MUGA
* No dyspnea at rest
* No exercise intolerance
* Oxygen saturation (SpO_2) > 94% by pulse oximetry (if there is a clinical indication for SpO_2 assessment)
* Not pregnant or nursing
* Negative pregnancy test
* No documented infection that is unresponsive to appropriate antibiotic, antiviral, or antifungal therapy
* No grade 2 or greater CNS toxicity
* Seizure disorder allowed if well controlled and on anticonvulsants
* See Disease Characteristics
* Recovered from prior immunotherapy
* At least 1 week since prior antineoplastic biologic agents
* Prior SCT allowed if the following criteria are met:

  * At least 60 days since prior SCT
  * Full hematopoietic reconstitution post-SCT
* No evidence of active acute or chronic graft-versus-host disease if post- allogeneic SCT
* No concurrent sargramostim (GM-CSF)
* See Disease Characteristics
* At least 3 weeks since prior myelosuppressive chemotherapy (4 weeks for nitrosourea) and recovered
* See Disease Characteristics
* Recovered from prior radiotherapy
* No concurrent medications that would interact with the study drug

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2002-06; Primary Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
MTD, defined as that dose at which fewer than one-third of patients experience DLT graded according to the NCI CTC v 2.0 | Up to day 49

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Cairo, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States